CLINICAL TRIAL: NCT02458105
Title: Acceptance & Commitment Therapy for Psychotic Inpatients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Required resources not available at the moment.
Sponsor: Uppsala University (Other)
Collaborators: Stockholm University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014/541
Record Dates: First submitted 2015-05-27; First posted 2015-05-29 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Acute Psychosis
Keywords: Acceptance and commitment therapy; Cognitive behavior therapy
MeSH Terms: interventions — Acceptance and Commitment Therapy; Neuropsychological Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acceptance & Commitment Therapy (Experimental): A variant of cognitive behavior therapy focused on acceptance and valued living in the presence of distressing symptoms.
  Interventions: Behavioral: Acceptance & Commitment Therapy
- Attention (Active Comparator): Supportive conversation at a frequency and length corresponding to the experimental condition.
  Interventions: Behavioral: Attention

INTERVENTIONS:
Behavioral: Acceptance & Commitment Therapy — A variant of cognitive behavior therapy focused on acceptance and valued living in the presence of distressing symptoms.
  Arms: Acceptance & Commitment Therapy
Behavioral: Attention — Supportive conversation at a frequency and length corresponding to the experimental condition.
  Arms: Attention

SUMMARY:
The overarching aim of the research project is to investigate whether Acceptance & Commitment Therapy (ACT) is an efficacious psychotherapeutic method of treatment for inpatients suffering from acute psychosis.

The method will be applied in two ways. Firstly, as an individual treatment for patients. Secondly, as an integrated part of the daily work on an inpatient ward, administered by nurses and assistant nurses trained in the method.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to a specified psychiatric inpatient ward during the time-period of the study; psychotic spectrum diagnosis as specified in patient charts; assessed by contact person on the ward as having delusions or hallucinations.

Exclusion Criteria:

* Cognitive difficulties to an extent where informed consent cannot be given.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-04; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Rehospitalization | 12 months
  Whether or not, and if so for how many days, a patient has ben readmitted to inpatient care during the follow-up period.

SECONDARY OUTCOMES:
Bull's Eye Values Inventory | 12 months
  Quality of life instrument to be administered before treatment, after treatment, and at 3, 6 and 12 month follow-up.
EQ-5D | 12 months
  Health related quality of life instrument to be administered before treatment, after treatment, and at 3, 6 and 12 month follow-up.
Clinical Global Impression Scale | 12 months
  Symptom severity instrument to be administered before treatment, after treatment, and at 3, 6 and 12 month follow-up.
Acceptance & Action Questionnaire | 12 months
  Psychological flexibility instrument to be administered before treatment, after treatment, and at 3, 6 and 12 month follow-up.
Psychotic Symptom Rating Scales | 12 months
  Symptom severity instrument to be administered before treatment, after treatment, and at 3, 6 and 12 month follow-up.
Checklist of Unit Behaviors | During inpatient care.
  Measure for degree of activity on the ward.

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Lundgren, PhD, Study Director — Stockholm University; Karolinska Institutet, department of Clinical Neuroscience & Centre for Psychiatry Research and Education, Stockholm County Council
Locations (1):
- Västmanland Hospital, Västerås, Västmanland County Council, Västerås, Sweden